CLINICAL TRIAL: NCT02616276
Title: Postprandial Effect of Breakfast Glycemic Index on Vascular Function, Insulinemia and Cognitive Performance, a Crossover Clinical Trial (BGI Study)
Brief Title: Postprandial Effect of Breakfast Glycemic Index on Vascular Function, Insulinemia and Cognitive Performance (BGI Study)
Acronym: BGI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion y Formacion en Ciencias de la Salud (Other)
Collaborators: Castilla-León Health Service (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: GRS 1192/B/15
Record Dates: First submitted 2015-11-19; First posted 2015-11-26 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Healthy
Keywords: Glycemic Index; Postprandial Period; Vascular Stiffness; Blood glucose; Cognition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Active Comparator): Control breakfast
  Interventions: Other: Control breakfast; Other: High glycemic index breakfast; Other: Low glycemic index breakfast
- Intervention 1 (Experimental): High glycemic index breakfast
  Interventions: Other: Control breakfast; Other: High glycemic index breakfast; Other: Low glycemic index breakfast
- Intervention 2 (Experimental): Low glycemic index breakfast
  Interventions: Other: Control breakfast; Other: High glycemic index breakfast; Other: Low glycemic index breakfast

INTERVENTIONS:
Other: Control breakfast — It consists of 350 ml of water at room temperature.
  Other Names: BF-1
Other: High glycemic index breakfast — It consists of 350 ml of water at room temperature, 200 ml of grape juice (with 136.28 kcal), 40 g of white bread (2 slices of 52.2 kcal each) and 29 g of strawberry jam (with 127.52 kcal); providing a total of 368.2 kcal.
  Other Names: BF-2
Other: Low glycemic index breakfast — It consists of 350 ml of water at room temperature, a 150 g apple (with 81.12 kcal), a 125 g low-fat natural yogurt (with 56.10 kcal), 3 shelled walnuts (with 38.94 kcal per unit) and 17.5 g of 72% black chocolate (with 102 kcal); supplying a total of 356.04 kcal.
  Other Names: BF-3

SUMMARY:
This is a crossover clinical trial aimed at adults (aged 20-40 years, with no cardiovascular disease), selected by consecutive sampling at urban primary care health clinics in Salamanca (Spain). Each subject will complete three interventions, with a washout period of one week: control breakfast (water), low glycemic index breakfast (apple, yogurt, walnuts and black chocolate) and high glycemic index breakfast (grape juice, bread and strawberry jam). The postprandial effect will be assessed at 60 and 120 minutes from each breakfast, measuring blood glucose and insulin and cognitive performance. Measurements will be performed of central blood pressure, augmentation index, pulse wave velocity, cardiac output and total peripheral vascular resistance at minutes (-10, 0, +15, +30, +45, +60, +75, +90, +105 and +120).

DETAILED DESCRIPTION:
Objectives:

The primary objective of this study is to evaluate the postprandial effect of low and high glycemic index breakfasts on vascular function, measured by central blood pressure, augmentation index and pulse wave velocity, in a sample of healthy young adults. The second objective is to assess the postprandial effect of low and high glycemic index breakfasts on blood glucose and insulin values in a sample of healthy young adults. The third and last objective is to assess the postprandial effect of low and high glycemic index breakfasts on cognitive performance in a sample of healthy young adults.

Design and setting:

A controlled crossover clinical trial, where each subject will complete three interventions (control breakfast, high glycemic index breakfast and low glycemic index breakfast), with a washout period of one week between each, and whose order will be determined by a randomization sequence generated using the Randomization.com software (http://www.randomization.com).

Study setting:

The study will be conducted in the primary care health area of Salamanca in the Research Unit of La Alamedilla, belonging to the Spanish Network for Preventive Activities and Health Promotion (redIAPP) and Salamanca Institute for Biomedical Research (IBSAL).

Study population:

The subjects of the study population will be selected by consecutive sampling in the primary care clinics of urban health centers in Salamanca (Spain) between 2015 and 2016. As this crossover clinical trial, a consecutive sampling will ensure comparability of the groups.

Intervention:

Each of the three scheduled visits will last approximately 2 and a half hours, and will be structured as follows:

Min -10: Measurement of clinical blood pressure, central blood pressure, and central hemodynamic parameters; evaluation of cognitive performance; laboratory test sampling to determine glucose and insulin blood levels.

Min 0: Measurement of central blood pressure and central hemodynamic parameters; intake of assigned breakfast (10 minutes).

Min +15, +30, +45: Measurement of central blood pressure and central hemodynamic parameters.

Min +60: Measurement of central blood pressure and central hemodynamic parameters; evaluation of cognitive performance; laboratory test sampling to determine glucose and insulin blood levels.

Min +75, +90, +105: Measurement of central blood pressure and central hemodynamic parameters.

Min +120: Measurement of central blood pressure and central hemodynamic parameters; evaluation of cognitive performance; laboratory test sampling to determine glucose and insulin blood levels.

ELIGIBILITY:
Inclusion Criteria:

* Young adults.
* Aged between 20 and 40 years.
* Both sexes.
* Those agree to sign the informed consent.

Exclusion Criteria:

* History of cardiovascular events (acute myocardial infarction, stroke, etc.).
* History of hypertension, diabetes mellitus or dyslipidemia.
* Pharmacological treatment for any of the above conditions.
* Diagnosis of clinically demonstrable neurological and/or neuropsychological disease.
* Excessive consumption of toxic substances.
* Celiac patients and/or those intolerant to lactose.
* Subjects on a low-calorie and/or low-sodium diet.
* Pregnant women.
* Those with any other circumstance that the investigators consider could interfere with the study procedures.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Augmentation index | Changes in augmentation index at 1 week, according to glycemic index of the breakfast
  Measurement by Mobil-O-Graph® device

SECONDARY OUTCOMES:
Central blood pressure | Changes in central blood pressure at 1 week, according to glycemic index of the breakfast
  Measurement by Mobil-O-Graph® device
Pulse wave velocity | Changes in pulse wave velocity at 1 week, according to glycemic index of the breakfast
  Measurement by Mobil-O-Graph® device
Blood glucose | Changes in blood glucose at 1 week, according to glycemic index of the breakfast
  Measurement by laboratory test sampling
Insulin values | Changes in insulin values at 1 week, according to glycemic index of the breakfast
  Measurement by laboratory test sampling
Immediate verbal memory | Changes in immediate verbal memory at 1 week, according to glycemic index of the breakfast
  Assessment by immediate recall of a list of 15 words, in three attempts
Delayed verbal memory | Changes in delayed verbal memory at 1 week, according to glycemic index of the breakfast
  Assessment by free recall of the words learnt in the first part of the study after a period of approximately 10 minutes
Phonological fluency | Changes in phonological fluency at 1 week, according to glycemic index of the breakfast
  Assessment by enumerating for one minute as many words as possible starting with different letters
Attention | Changes in attention at 1 week, according to glycemic index of the breakfast
  Assessment by Trail Making Test A
Processing speed | Changes in processing speed at 1 week, according to glycemic index of the breakfast
  Assessment by Trail Making Test B
Executive functions | Changes in executive functions at 1 week, according to glycemic index of the breakfast
  Assessment by Trail Making Test B
Working memory | Changes in working memory at 1 week, according to glycemic index of the breakfast
  Assessment by WAIS Digit Span Backward test
Sustained attention | Changes in sustained attention at 1 week, according to glycemic index of the breakfast
  Assessment by Stroop test
Selective attention | Changes in selective attention at 1 week, according to glycemic index of the breakfast
  Assessment by Stroop test

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Care Research Unit - The Alamedilla Center for Health, Salamanca, Salamanca, Spain

REFERENCES:
- [Derived] Sanchez-Aguadero N, Garcia-Ortiz L, Patino-Alonso MC, Mora-Simon S, Gomez-Marcos MA, Alonso-Dominguez R, Sanchez-Salgado B, Recio-Rodriguez JI. Postprandial effect of breakfast glycaemic index on vascular function, glycaemic control and cognitive performance (BGI study): study protocol for a randomised crossover trial. Trials. 2016 Oct 24;17(1):516. doi: 10.1186/s13063-016-1649-x. PMID 27776536